CLINICAL TRIAL: NCT07125703
Title: Observational Study With Additional Procedures: Metabolomic and Ultrastructural Findings of Allograft in Heart Transplantation and Their Correlation With Graft Dysfunction.
Acronym: MetabolHeart
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefano Pelenghi, Stefano Pelenghi, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: MetabolHeart
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-02

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This is a single center retrospective/prospective observational study with additional procedures meant to evaluate molecular mechanisms underlying injury in donor's heart.

The research project will focus on Metabolomics by NMR and LC-MS and ultrastructural analysis using electron microscopy of endomyocardial biopsies (EMB).In our clinical protocol of heart transplantation, myocardial biopsy samples are routinely provided at intraoperative and postoperative time.

ELIGIBILITY:
Inclusion Criteria:

- Informed Consent available

Exclusion Criteria:

* Uncomplete donor data collection
* Patients undergoing heart-lung bloc transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially all patients undergoing heart transplant at the Cardiac Surgery - Fondazione IRCCS Policlinico San Matteo, Pavia until 31-12-2024
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biventricular failure: left ventricular failure (LV EF <40%) and right ventricular failure (TAPSE <16% and/or FAC < 35% and/or S' wave velocity < 10 cm/sec) within 24 hours post transplantation | Within 24 hours post transplantation

SECONDARY OUTCOMES:
Left ventricular dysfunction (longitudinal global strain (LGS) < -14% at 1 month and <-17% at 6 and 12 months and/or FEvsx <50%) at 1, 6, 12 months after transplant (in absence of rejection) | At 1, 6, 12 months after transplant
Left ventricular failure (LV EF <40%) within 24 hours post transplantation | Within 24 hours post transplantation
Right ventricular failure (TAPSE <16% and/or FAC < 35% and/or S' wave velocity < 10 cm/sec) within 24 hours post transplantation | Within 24 hours post transplantation
Hemodynamic: Cardiac Index < 2 L/min/mq, wedge pressure >20 mmHg, right atrial pressure (RAP > 15 mmHg) within 24 hours post transplantation and at 1, 6, 12 months after transplant (in absence of rejection) | At 1, 6, 12 months after transplant
Death for graft failure within 24 hours post transplantation | Within 24 hours post transplantation
ECMO within 24 hours of transplant for ventricular failure | Within 24 hours of transplant
IABP within 24 hours of transplant for ventricular failure | Within 24 hours of transplant
Echocardiographic parameters: E/A>>1; DT<150 msec; E/e'>15, atrial strain at 1, 6, 12 months after transplant (in absence of rejection) | At 1, 6, 12 months after transplant
Death at 1, 6, 12 months after transplant (in absence of rejection | At 1, 6, 12 months after transplant
Trend of cardiac biomarker (BNP), trend of TNIhs, angiotensinogen, ADIPOQ, HGFAC, IGFBP3, other markers of ischaemia | At first and third week

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy